CLINICAL TRIAL: NCT02613104
Title: Emotion Recognition Modification for Bipolar Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Anna Van Meter, Assistant Professor, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-2811
Record Dates: First submitted 2015-11-18; First posted 2015-11-24 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sad to Happy (Experimental): emotion recognition modification - sad>happy
  Interventions: Other: emotion recognition modification - sad>happy
- Sad control (Placebo Comparator): emotion recognition modification - sad>happy control
  Interventions: Other: emotion recognition modification - sad>happy control
- Angry to Happy (Experimental): emotion recognition modification - angry>happy
  Interventions: Other: emotion recognition modification - angry>happy
- Angry control (Placebo Comparator): emotion recognition modification - angry>happy control
  Interventions: Other: emotion recognition modification - angry>happy control

INTERVENTIONS:
Other: emotion recognition modification - sad>happy — Participants must choose whether each face is happy or sad. Based on these responses, an algorithm then estimates each participant's balance point, the threshold point on the morph sequence at which they are equally likely to label the face as happy or sad. During the intervention, the participant receives feedback on their emotion choices designed to train them to identify two additional morphs as happy, rather than sad. The intervention is completed three times.
  Arms: Sad to Happy
Other: emotion recognition modification - sad>happy control — Participants must choose whether each face is happy or sad. Based on these responses, an algorithm then estimates each participant's balance point, the threshold point on the morph sequence at which they are equally likely to label the face as happy or sad. During the placebo intervention, the participant receives feedback on their emotion choices designed to reinforce their initial emotion choices. The placebo intervention is completed three times.
  Arms: Sad control
Other: emotion recognition modification - angry>happy — Participants must choose whether each face is happy or angry. Based on these responses, an algorithm then estimates each participant's balance point, the threshold point on the morph sequence at which they are equally likely to label the face as happy or angry. During the intervention, the participant receives feedback on their emotion choices designed to train them to identify two additional morphs as happy, rather than angry. The intervention is completed three times.
  Arms: Angry to Happy
Other: emotion recognition modification - angry>happy control — Participants must choose whether each face is happy or angry. Based on these responses, an algorithm then estimates each participant's balance point, the threshold point on the morph sequence at which they are equally likely to label the face as happy or angry. During the placebo intervention, the participant receives feedback on their emotion choices designed to reinforce their initial emotion choices. The placebo intervention is completed three times.
  Arms: Angry control

SUMMARY:
Previous research suggests that people with bipolar disorder have trouble accurately identifying emotions. The goal of this study is to test a novel intervention, emotion recognition modification (ERM), to help improve the ability of young people with bipolar disorder to identify emotions.

DETAILED DESCRIPTION:
Procedure: Participants will be recruited through the University Clinic, affiliated psychiatric hospitals and outpatient psychiatric clinics in the area, and public websites. Interested participants will be interviewed on the phone to determine initial eligibility; those who meet criteria will be invited for a comprehensive evaluation.

For potential participants under the age of 18, parents/caregivers will be asked the eligibility questions about their child. If the child meets initial eligibility criteria, both s/he and the parent/caregiver will be invited to the baseline appointment.

The baseline appointment will take place at Zucker Hillside Hospital. Following the informed consent/assent process, participants will be interviewed by a trained research assistant to assess clinical and treatment history, and to determine diagnostic eligibility, using the SCID. Participants who meet eligibility criteria will proceed to complete other baseline measures.

Emotion recognition baseline procedure. The baseline task allows for the measurement of each participants' baseline balance point, the point at which they are equally likely to see a given face as happy or sad (or angry). Each participant will complete 45 trials of the emotion recognition task in which each face from a morph sequence of happy and sad (or angry) faces is presented, the participant is then forced to decide whether a face is sad (or angry) or happy.

Intervention: Once the baseline measures are completed, participants will be randomized to the sad-to-happy condition, the angry-to-happy condition, or a control condition (n =20 per group). Participants in the intervention conditions will complete the training task three times over three in-person sessions. The task will be similar to the baseline procedure; participants will view faces and be asked to judge the expression, however they will now be given feedback (e.g. "Incorrect! That face was happy."), in order to shift the category of happy faces to include those faces two morph steps beyond the participant's baseline balance point. Participants in the control condition will repeat the baseline task, with feedback consistent with their baseline performance (i.e. the faces they judged as happy initially will be called "correct" when judged happy again. The intervention will be administered a total of three times (once at baseline, once at the first follow-up, once at the second follow-up).

Follow-Up: After the final training session, participants will complete the first follow-up. This will consist of the clinician-administered YMRS, as well as online questionnaires, including the LEE, PANAS, GBI, social network task, Perceived Social Support, feasibility questionnaire.

Eight weeks after completing the final training session, participants will return to the research lab for the final follow-up, which will include the following measures, LEE, PANAS, GBI, social network task, Perceived Social Support, emotion recognition task, YMRS, and BDI-II to assess changes in mood episode over the study follow-up period. Participants will also be asked to complete a brief form about whether they liked the intervention and found it convenient to assess burden and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-25 with a bipolar spectrum disorder. Must be English-speaking.

Exclusion Criteria:

* Participants who have cognitive impairment, current psychosis, current suicidal intent, or current substance use disorder will be excluded.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
change in face emotion recognition as assessed by the number of face emotions correctly identified | two months after the completion of the intervention
  Ratio of faces identified as happy versus sad/angry

SECONDARY OUTCOMES:
change in self reported depressed mood as measured by baseline and post intervention | following three sessions of the intervention (approximately two weeks)
  General Behavior Inventory
change in clinician-rated depressed mood as measured by baseline and post intervention scores o | following three sessions of the intervention (approximately two weeks)
  Beck Depression Inventory
change in self-reported depressed mood as measured by baseline and two month follow-up scores | two months after completion of intervention
  General Behavior Inventory
change in clinician-rated depressed mood as measured by baseline and two month follow-up scores | two months after completion of intervention
  Beck Depression Inventory
change in social functioning as measured by the social network questionnaire | following three sessions of the intervention (approximately two weeks)
  Social network questionnaire
change in social functioning as measured by the social network questionnaire at follow-up | two months after completion of intervention
  Social network questionnaire
change in positive affect as measured by the Positive and Negative Affect Scale | following three sessions of the intervention (approximately two weeks)
  PANAS
change in positive affect as measured by the Positive and Negative Affect Scale at follow-up | two months after completion of intervention
  PANAS

CONTACTS AND LOCATIONS:
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

REFERENCES:
- [Background] Penton-Voak IS, Bate H, Lewis G, Munafo MR. Effects of emotion perception training on mood in undergraduate students: randomised controlled trial. Br J Psychiatry. 2012 Jul;201(1):71-2. doi: 10.1192/bjp.bp.111.107086. Epub 2012 Apr 26. PMID 22539781
- [Background] Penton-Voak IS, Thomas J, Gage SH, McMurran M, McDonald S, Munafo MR. Increasing recognition of happiness in ambiguous facial expressions reduces anger and aggressive behavior. Psychol Sci. 2013 May;24(5):688-97. doi: 10.1177/0956797612459657. Epub 2013 Mar 26. PMID 23531485